CLINICAL TRIAL: NCT02584088
Title: Ultrasound Appearance of the Endometrium Post Radio-Frequency Ablation
Status: Completed | Type: Observational
Sponsor: TriHealth Inc. (Other)
Responsible Party: Sponsor
Other Study IDs: 15-029
Record Dates: First submitted 2015-10-20; First posted 2015-10-22 (Estimated); Last update posted 2022-12-02 (Actual); Status verified 2022-12

CONDITIONS: Menorrhagia
Keywords: NovaSure; Ablation; Menorrhagia; Endometrium
MeSH Terms: conditions — Menorrhagia | interventions — High-Energy Shock Waves

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: Ultrasound — The appearance of the post ablative endometrium on transvaginal ultrasound at 2, 6, and 12 months.

SUMMARY:
* The study primarily aims to evaluate the post ablative endometrium and uterus using transvaginal ultrasound to provide descriptive information as to what may be expected in the 12 months after a NovaSure ablation. Investigators believe this knowledge will help them to determine when to proceed with further evaluation postoperatively or when to counsel patients on expectant management based on ultrasonographic findings.
* Secondary aims include correlation of ultrasonographic findings to demographic patient data.

DETAILED DESCRIPTION:
Heavy and irregular menses affects 9-14% of gynecologic patients. Surgical can be employed intervention is sought when medical management fails. Endometrial ablation or desiccation of the endometrium using minimally invasive instruments has been utilized in this scenario. The current mainstay intervention is non-resectoscopic radio frequency ablation. These procedures have high satisfaction rates (81 to 93%) similar to hysterectomy and leave up to 47% of patients amenorrheic. Post operative complications, both short and long term, and failure rates have been well studied. A limited number of studies have been performed to assess the histologic state of the post ablative endometrium and fewer assessing the radiographic appearance of the endometrium. Therefore, this current study aims to describe the ultrasonographic appearance of the post ablative endometrium and uterus.

ELIGIBILITY:
Inclusion Criteria:

* women of premenopausal age
* 18 years and older
* intended ablative management of menorrhagia

Exclusion Criteria:

* uterine cavity anatomic abnormality
* previous uterine ablation procedure
* previous cervical procedure
* presence of submucosal fibroids
* tissue diagnosis of endometrial hyperplasia/endometrial carcinoma
* pregnancy and delivery less than 1 year before ablation.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients who are candidates for NovaSure ablation for treatment of menorrhagia.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2016-10-11 (Actual); Primary Completion 2021-11 (Actual); Study Completion 2021-11 (Actual)

PRIMARY OUTCOMES:
Endometrial thickness (measured using a scale) | 2 months

CONTACTS AND LOCATIONS:
Overall Officials: Catrina Crisp, MD, MSc, Principal Investigator — TriHealth Inc.
Locations (2):
- United States (2):
  - Good Samaritan Hospital, Cincinnati, Ohio
  - Bethesda North Hospital, Cincinnati, Ohio

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] El-Nashar SA, Hopkins MR, Creedon DJ, St Sauver JL, Weaver AL, McGree ME, Cliby WA, Famuyide AO. Prediction of treatment outcomes after global endometrial ablation. Obstet Gynecol. 2009 Jan;113(1):97-106. doi: 10.1097/AOG.0b013e31818f5a8d. PMID 19104365
- [Background] Dickersin K, Munro MG, Clark M, Langenberg P, Scherer R, Frick K, Zhu Q, Hallock L, Nichols J, Yalcinkaya TM; Surgical Treatments Outcomes Project for Dysfunctional Uterine Bleeding (STOP-DUB) Research Group. Hysterectomy compared with endometrial ablation for dysfunctional uterine bleeding: a randomized controlled trial. Obstet Gynecol. 2007 Dec;110(6):1279-89. doi: 10.1097/01.AOG.0000292083.97478.38. PMID 18055721
- [Background] Alhilli MM, Wall DJ, Brown DL, Weaver AL, Hopkins MR, Famuyide AO. Uterine ultrasound findings after radiofrequency endometrial ablation: correlation with symptoms. Ultrasound Q. 2012 Dec;28(4):261-8. doi: 10.1097/RUQ.0b013e318276653b. PMID 23149510
- [Background] Ahonkallio SJ, Liakka AK, Martikainen HK, Santala MJ. Feasibility of endometrial assessment after thermal ablation. Eur J Obstet Gynecol Reprod Biol. 2009 Nov;147(1):69-71. doi: 10.1016/j.ejogrb.2009.06.014. Epub 2009 Jul 16. PMID 19615812
- [Background] Penninx JPM, Herman MC, Mol BW, Bongers MY. Five-year follow-up after comparing bipolar endometrial ablation with hydrothermablation for menorrhagia. Obstet Gynecol. 2011 Dec;118(6):1287-1292. doi: 10.1097/AOG.0b013e318236f7ed. PMID 22105257
- [Background] Luo X, Lim CE, Li L, Wong WS. Hysteroscopic appearance of endometrial cavity after microwave endometrial ablation. J Minim Invasive Gynecol. 2010 Jan-Feb;17(1):30-6. doi: 10.1016/j.jmig.2009.09.012. PMID 20129329
- [Background] Onoglu A, Taskin O, Inal M, Sadik S, Simsek M, Akar M, Kursun S, Mendilcioglu I, Postaci H, Ispahi C. Comparison of the long-term histopathologic and morphologic changes after endometrial rollerball ablation and resection: a prospective randomized trial. J Minim Invasive Gynecol. 2007 Jan-Feb;14(1):39-42. doi: 10.1016/j.jmig.2006.06.027. PMID 17218227
- [Background] Taskin O, Onoglu A, Inal M, Turan E, Sadik S, Vardar E, Postaci H, Wheeler JM. Long-term histopathologic and morphologic changes after thermal endometrial ablation. J Am Assoc Gynecol Laparosc. 2002 May;9(2):186-90. doi: 10.1016/s1074-3804(05)60130-2. PMID 11960046
- [Background] Leung PL, Tam WH, Yuen PM. Hysteroscopic appearance of the endometrial cavity following thermal balloon endometrial ablation. Fertil Steril. 2003 May;79(5):1226-8. doi: 10.1016/s0015-0282(02)04956-7. PMID 12738523
- [Background] Colgan TJ, Shah R, Leyland N. Post-hysteroscopic ablation reaction: a histopathologic study of the effects of electrosurgical ablation. Int J Gynecol Pathol. 1999 Oct;18(4):325-31. doi: 10.1097/00004347-199910000-00006. PMID 10542940